CLINICAL TRIAL: NCT02749201
Title: Transmitted Light Tissue Thickness Analysis (TiLTT)
Acronym: TiLLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Danny A Sherwinter, Chief Minimally Invasive Surgery, Maimonides Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-06-15-MMC
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Morbid Obesity
Keywords: Obesity; sleeve gastrectomy
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Analysis (Experimental): Light Intensity and gastric wall thickness analysis
  Interventions: Device: Gastrisail

INTERVENTIONS:
Device: Gastrisail — Light Intensity and gastric wall thickness assessment

SUMMARY:
To assess gastric wall thickness using transmitted light intensity.

DETAILED DESCRIPTION:
The most common surgical procedure for weight loss is the sleeve gastrectomy. The laparoscopic sleeve gastrectomy (LSG) involves the linear stapling of the stomach using a stapling device [e.g. Echelon (Ethicon Somerset NJ)] fired multiple times along the length of the stomach thereby excising 80-90% of the stomach leaving the patient with a "sleeve" of stomach rather than the normal anatomical pouch. The gastric wall varies in thickness and thus there are a varied staple sizes available for this use. Staple sizes range from 2.0mm-5.0mm in height. In standard surgical practice the surgeon chooses the size of staple cartridge for each subsequent firing based on his experience and estimations about the thickness of the stomach tissue in any given region. The drawback of this technique is that it is highly inaccurate. If the surgeon's estimation is in error, the staple height chosen may be either too tall or too short leading to bleeding or leakage from between the staples or malformed/unformed staples leading to staple line failure. Any of these errors can lead to devastating complications such as hemorrhage, leak, sepsis and death. To date there is no objective way to measure the thickness of the tissue being stapled and thus staple choice relies entirely on surgeon estimation which is inherently inaccurate. The investigators hypothesize that a light source placed in the stomach lumen will transmit light through the gastric wall. The amount of light transmitted, i.e. visible to an imaging device arrayed external to the stomach, will be directly proportionate to the thickness of the stomach. This study will take advantage of the fact that during routine procedures in the sleeve gastrectomy procedure a lighted tube is placed into the gastric lumen via the mouth. This device is called the Gastrisail and has 10 separate LED lights arrayed along its length. This allows for the measurement of transmitted light intensity through the gastric wall at 10 individual locations along the length f the stomach. In addition this study will take advantage of the fact that during standard practice in a sleeve gastrectomy a section of the stomach corresponding to the location of the lights is excised and sent for pathological evaluation. This will allow us to measure the actual thickness of the stomach at 10 points corresponding to he locations of the transmitted light intensity. For this measurement The investigators will use a standardized and validated measurement tool/calipers. Now with two sets of numbers the investigators plan to correlate the degree of transmitted light intensity with actual thickness measurements and thereby reach an algorithm which will allow the transmitted light intensity data alone to predict gastric wall thickness. This will provide the surgeon with an entirely non-invasive objective measure of gastric wall thickness and hopefully improve his/her choice of staple size during these surgical procedures thus improving safety.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent
* Subject is between the ages of 18 and 80 years of age
* Subject is scheduled for and undergoes primary sleeve gastrectomy

Exclusion Criteria:

* Revisional Bariatric Surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Sherwinter, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Analysis
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Analysis
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Transmitted Light Intensity to Gastric Wall Thickness)
Description: Number of patients with transmitted light intensity to gastric wall thickness between the groups
Time Frame: intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: Intraoperative only
Arm/Group | Analysis
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT02749201/Prot_SAP_000.pdf